CLINICAL TRIAL: NCT01083147
Title: Age-Related Macular Degeneration (AMD) - Beta Study Telemedicine Assessment
Acronym: AMD
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Osnat Ehrman/Clinical manager, Notal Vision
Organization: Notal Vision Inc. (Industry)
Other Study IDs: ForeseeHome-US3
Record Dates: First submitted 2010-03-07; First posted 2010-03-09 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Age-Related Macular Degeneration
Keywords: Intermediate AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dry AMD: subjects diagnosed as intermediate AMD in at least one eye
  Interventions: Device: FORESEE HOME

INTERVENTIONS:
Device: FORESEE HOME — Home Monitoring

SUMMARY:
The purpose of this study is to evaluate the compliance of the Foresee Home device in intermediate AMD patients.

DETAILED DESCRIPTION:
This is a non-randomized cohort, multi-center study. The eligible subjects will be asked to use the FORESEE HOME device daily and the tests results will be automatically transmitted to the Data Monitor Center for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who successfully completed participation in ForeseeHome-US2 study
* Patients with ability to comprehend and sign the informed consent/authorization

Exclusion Criteria:

* Subjects who failed to complete participation in ForeseeHome-US2 study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intermediate AMD
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Subject compliance with Foresee HomeTM device | 6 months

SECONDARY OUTCOMES:
Assessment of the Telemedicine infrastructure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roth, MD, Principal Investigator — Vitreos retina center - NJ
Locations (1):
- Vitreos retina center, Toms River, New Jersey, United States